CLINICAL TRIAL: NCT02502929
Title: Lifestyle and Medication Management to Lower Diabetes Risk in Severe Mental Illness
Brief Title: Diabetes Risk Reduction Through Eat, Walk, Sleep and Medication Therapy Management for Depressed Cambodians
Acronym: DREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Khmer Health Advocates (Unknown); Penn State University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Julie A. Wagner, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-164S-3; 5R01DK103663 (NIH)
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Diabetes; Depression
Keywords: Diabetes; Depression; Medication therapy management; Community health workers; Cambodian; Refugee; Prevention
MeSH Terms: conditions — Diabetes Mellitus; Depression | interventions — Social Work; Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Social Services (Active Comparator): Participants in this arm will receive referrals for social services as indicated.
  Interventions: Behavioral: Social Services
- Lifestyle (Experimental): Participants in this arm will receive lifestyle modification from community health workers using the manualized lifestyle intervention called "Eat, Walk, Sleep". They will receive individual home visits, health activity group sessions, and supportive phone calls.
  Interventions: Behavioral: Lifestyle
- Lifestyle plus Medication Therapy Management (Experimental): Participants in this arm will receive everything in the Lifestyle arm, plus Medication Therapy Management (MTM). Participants will receive MTM from a pharmacist via telemedicine with the assistance of a community health worker.
  Interventions: Behavioral: Lifestyle Plus Medication Therapy Management

INTERVENTIONS:
Behavioral: Social Services
  Arms: Social Services
Behavioral: Lifestyle
  Arms: Lifestyle
Behavioral: Lifestyle Plus Medication Therapy Management
  Arms: Lifestyle plus Medication Therapy Management

SUMMARY:
The primary aim of the study is to compare the effect of three different interventions on lifestyle risk factors and biological risk factors for type 2 diabetes in depressed Cambodians. The three different interventions are lifestyle, lifestyle plus medication therapy management, and social services.

DETAILED DESCRIPTION:
Cambodian Americans have high risk for major depressive disorder and for type 2 diabetes. Depression is a known risk factor for diabetes. Some antidepressants can also increase risk of diabetes by causing weight gain. DREAM will test the effect of lifestyle and medication therapy management (MTM) compared to social services (control) on diabetes risk among depressed Cambodian Americans. Community health workers (CHWs) will deliver the lifestyle intervention and assist pharmacists with MTM. Lifestyle and biological risk factors for diabetes, such as depressive symptoms, HbA1c and insulin sensitivity, will be measured before and after the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as Cambodian or Cambodian-American
* Khmer speaking
* Likely major depressive disorder
* Elevated diabetes risk score per ADA guidelines
* Ambulatory
* Competent to give consent.

Exclusion Criteria:

* Pregnancy or plans to become pregnant in the next 2 years
* Previous diagnosis of diabetes
* Seeing or hearing problems that would interfere with group sessions
* Currently being followed by a physician for major medical problem
* Serious thinking or memory problems (e.g., schizophrenia or dementia)
* 3 or more days in a psychiatric hospital or self-harm in the past 2 years.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Lifestyle risk for type 2 diabetes | 12 months and 15 months
  Change from baseline in depressive symptoms according to the Hopkins Symptom Checklist
Biological risk for type 2 diabetes | 12 months and 15 months
  Change from baseline in HbA1c and insulin resistance according to logHOMA-IR

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Wagner, PhD, Principal Investigator — UConn Health
Locations (3):
- United States (3):
  - Uconn Health, Farmington, Connecticut
  - Khmer Health Advocates, West Hartford, Connecticut
  - Center for Southeast Asians, Providence, Rhode Island

REFERENCES:
- [Derived] Wagner JA, Bermudez-Millan A, Buckley TE, Buxton OM, Feinn RS, Kong S, Kuoch T, Master L, Scully MF. Secondary analysis of a randomized trial testing community health educator interventions for diabetes prevention among refugees with depression: effects on nutrition, physical activity and sleep. Int J Behav Nutr Phys Act. 2023 Sep 12;20(1):107. doi: 10.1186/s12966-023-01509-y. PMID 37700288
- [Derived] Wagner J, Bermudez-Millan A, Buckley T, Buxton OM, Feinn R, Kong S, Kuoch T, Nye LM, Scully M. Self-reported outcomes of a randomized trial comparing three community health worker interventions for diabetes prevention among Cambodian Americans with depression. Patient Educ Couns. 2022 Dec;105(12):3501-3508. doi: 10.1016/j.pec.2022.09.011. Epub 2022 Oct 6. PMID 36307274
- [Derived] Wagner JA, Bermudez-Millan A, Berthold SM, Buckley T, Buxton OM, Feinn R, Kuoch T, Kong S, Lim M, Polomoff C, Scully M. Risk factors for drug therapy problems among Cambodian Americans with complex needs: a cross-sectional, observational study. Health Psychol Behav Med. 2022 Jan 24;10(1):145-159. doi: 10.1080/21642850.2021.2021917. eCollection 2022. PMID 35087696
- [Derived] Wagner J, Bermudez-Millan A, Buckley T, Buxton OM, Feinn R, Kong S, Kuoch T, Nahmod NG, Scully M. A randomized trial to decrease risk for diabetes among Cambodian Americans with depression: Intervention development, baseline characteristics and process outcomes. Contemp Clin Trials. 2021 Jul;106:106427. doi: 10.1016/j.cct.2021.106427. Epub 2021 May 3. PMID 33957272